CLINICAL TRIAL: NCT00962143
Title: Prospective, Randomized, Multi-center: Acute Achilles Repair With or Without OrthADAPT Augmentation
Brief Title: Acute Achilles Repair With or Without OrthADAPT Augmentation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Synovis Surgical Innovations (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: P07-044-CR
Record Dates: First submitted 2009-08-17; First posted 2009-08-19 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Achilles Tendon Tear
Keywords: Acute Achilles Tendon Tear; Acute Achilles Tendon Repair

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Achilles repair without OrthADAPT Augmentation (Active Comparator): Achilles repair without OrthADAPT Augmentation
  Interventions: Procedure: Achilles repair without OrthADAPT Augmentation
- Achilles repair with OrthADAPT augmentation (Experimental): Achilles repair with OrthADAPT augmentation
  Interventions: Device: Achilles repair with OrthADAPT augmentation

INTERVENTIONS:
Device: Achilles repair with OrthADAPT augmentation — Achilles repair with OrthADAPT augmentation
  Arms: Achilles repair with OrthADAPT augmentation
Procedure: Achilles repair without OrthADAPT Augmentation — Achilles repair without OrthADAPT Augmentation
  Arms: Achilles repair without OrthADAPT Augmentation

SUMMARY:
The purpose of this study is to assess the clinical performance of the OrthADAPT Bioimplant in patients with acute mid-substance Achilles tendon tears requiring surgical repair.

ELIGIBILITY:
Inclusion Criteria:

* A transverse, full thickness, acute mid-substance Achilles tendon tear that requires surgical repair
* Achilles tendon tear is repairable by surgery using primary means as determined by intra-operative assessment
* Achilles tendon rupture with viable ends of the tendon that are suitable for primary repair
* Isolated Achilles tendon rupture without poly trauma
* Patient must be 18 to 70 years of age
* Life expectancy greater than or equal to 12 months
* Patient is able to provide voluntary informed consent
* Patient is willing and able to return for all follow-up visits and study related exams
* Patient is willing to comply with prescribed physical therapy regimen

Exclusion Criteria:

* Emergency, poly trauma patients
* Previous Achilles tendon surgical procedure on that tendon
* Deficit in the contralateral extremity that prevents a comparison with the treated extremity
* Repair requires tendon lengthening, gap filling or tendon transfer
* BMI greater than 40
* Peripheral arterial disease
* Uncontrolled Diabetes Mellitis
* Patients whose injury is known to involve litigation
* Known allergy to equine derived product
* Systemic collagen disease
* Neurological disease
* Active infection - systemic or at the intended surgical site
* Acute use of immunosuppressive agents
* Rupture resulting from fluoroquinolone induced tendinopathy
* Alcohol or drug abuse
* Participant in another investigational drug or device trial
* Pathologic soft tissue conditions that would prevent secure surgical fixation
* Patients who are unwilling or unable to return for follow-up visits and study related exams
* Pregnant women
* Cancer patients
* Decisionally impaired patients
* Institutionalized patients
* Prisoners

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in ROM and Biodex Isokinetic Strength Testing compared to contralateral limb | 2, 3, 4.5, 6, and 12 months
Time to return to weight bearing | 2, 3, 4.5, 6, and 12 months
Time to return to full activity | 2, 3, 4.5, 6, and 12 months

SECONDARY OUTCOMES:
Swelling, stiffness, pain, disease specific quality of life: SF-36, AOFAS Hindfoot scores | 6 weeks, 2, 3, 4.5, 6 and 12 months
Complication rate including re-rupture and incision wound healing delay | 6 weeks, 2, 3, 4.5, 6 and 12 months
Incidence of device and procedure-related adverse events | 6 weeks, 2, 3, 4.5, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lee, DPM, Principal Investigator — Department of Orthopaedic Surgery, UCSD
Locations (1):
- Orthopaedic Institute of Central Jersey, Sea Girt, New Jersey, United States